CLINICAL TRIAL: NCT01081886
Title: A Prospective, Randomized, Controlled Superiority Study to Evaluate Use of the PEAK PlasmaBlade 4.0 in Total Knee Replacement
Brief Title: PEAK PlasmaBlade 4.0 Versus Traditional Electrosurgery in Total Knee Replacement.
Acronym: PRECISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination due to acquisition of PEAK Surgical by Medtronic
Sponsor: Medtronic Surgical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEAK VP-00082
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Degenerative Joint Disease; Osteoarthritis
Keywords: Total knee arthroplasty; PlasmaBlade; Electrosurgery; PEAK Surgical; Medtronic Advanced Energy; Medtronic
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Hyperthermia | interventions — Methods; Electrosurgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PlasmaBlade (Experimental): The PEAK PlasmaBlade will be used for the entirety of the total knee replacement, including the skin incision.
  Interventions: Device: PEAK PlasmaBlade 4.0
- Standard of Care (Active Comparator): Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
  Interventions: Device: Traditional Electrosurgery with scalpel

INTERVENTIONS:
Device: PEAK PlasmaBlade 4.0 — The PEAK PlasmaBlade will be used for the entirety of the total knee replacement, including the skin incision.
  Other Names: Intervention; PlasmaBlade
  Arms: PlasmaBlade
Device: Traditional Electrosurgery with scalpel — Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
  Other Names: Scalpel and electrosurgery; SOC
  Arms: Standard of Care

SUMMARY:
The objective of this clinical study is to evaluate the operative performance of the PEAK PlasmaBlade 4.0 during total knee replacement; to monitor and record post-operative pain, activity level, narcotic consumption, adverse events, and skin scarring following surgery; and compare these outcomes to the current standard of care (SOC).

DETAILED DESCRIPTION:
Total knee replacement is a surgical procedure performed to replace the weight-bearing surfaces of the knee joint. The goal of total knee replacement is to improve a patient's mobility by improving the function of the the knee joint.

The PEAK PlasmaBlade® uses pulsed radiofrequency (RF) energy and a highly-insulated handpiece design to enable precision cutting and coagulation at the point of application. The PlasmaBlade has received FDA clearance for use in plastic, general, orthopedic, and ear, nose, and throat (ENT) surgery, and has demonstrated a significantly reduced thermal injury profile in incised tissue compared to traditional electrosurgical devices. It is hypothesized that this benefit may improve the post-operative outcome of patients undergoing total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 and 80 years old
2. Physically healthy, stable weight
3. Requiring unilateral total knee arthroplasty (TKA)
4. Subject exhibits preoperative radiographic evidence of joint degeneration consistent with TKA that cannot be treated in non-operative fashion
5. Subject has severe knee pain and disability due to degenerative joint disease
6. Subject must understand the nature of the procedure and provide written informed consent prior to the procedure.
7. Subject must be willing and able to comply with all follow-up evaluations
8. Subject must be willing to undergo TKA using the Signature Knee System

Exclusion Criteria:

1. Age younger than 21 or greater than 80 years old
2. Previous history of infection in the affected joint
3. Peripheral vascular disease
4. Revision procedures
5. BMI > 35
6. Valgus or varus deformity > 15 degrees
7. Flexion contracture > 15 degrees
8. History of diabetes
9. Anticoagulation therapy which cannot be discontinued
10. Cognitive impairment or mental illness
11. Severe cardiopulmonary deficiencies
12. Known coagulopathy
13. Immunocompromised
14. Kidney disease (any type)
15. Unable to follow instructions or complete follow-up
16. Currently taking any medication known to affect healing
17. Currently enrolled in another investigational device or drug trial

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - DeClaire Knee and Orthopedic Institute, Rochester Hills, Michigan
  - Texas Health Arlington Memorial Hospital, Arlington, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SOC): Scalpel will be used for the skin incision and traditional electrosurgery for the subcutaneous dissection.
Period: Overall Study
Arm/Group | PlasmaBlade | Standard of Care (SOC)
Started | 11 | 13
Completed | 0 | 0
Not Completed | 11 | 13
Not completed — Study termination | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PlasmaBlade | Standard of Care (SOC) | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Customized [Number; unit: participants] — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. The protocol-specified age range is used for this baseline measure.
  participants
    21 to 80 years | 11 | 13 | 24
Gender [Number; unit: participants]
  Female | NA — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. | NA — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. | 0
  Male | NA — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. | NA — An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation. | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain
Description: Wong-Baker FACES Visual Analog Scale, 0 (no hurt) to 10 (hurts worst). The results represent the mean of each subject's mean pain scores over 10 days.
Time Frame: Postoperative (0 to 10 days)
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Operative Metrics: Operative Time, Estimated Blood Loss, Skin Scarring, Knee Society Score (KSS)
Time Frame: Intraoperatively and 1-2 weeks postoperatively
Population: An integrity audit found that the data for this study could not be analyzed owing to unverifiable source documentation.
Arm/Group | PlasmaBlade | Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | PlasmaBlade | Standard of Care (SOC)
Serious Adverse Events (participants affected / at risk) | 3/11 | 1/13
Other Adverse Events (participants affected / at risk) | 10/11 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PlasmaBlade (N=11) | Standard of Care (SOC) (N=13)
Spider bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PlasmaBlade (N=11) | Standard of Care (SOC) (N=13)
Insomnia (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain/swelling (Surgical and medical procedures) | 6 (8) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Effusion (Surgical and medical procedures) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Upon Medtronic's acquisition of PEAK surgical, a study integrity audit was undertaken. Results of the audit showed that patient's rights and safety were maintained, but the source data, including baseline demographics, were unverifiable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less